CLINICAL TRIAL: NCT02907333
Title: Use of Condoms in Prevention of Progression of Cervical Intraepithelial Neoplasia: A Randomized Controlled Trial.
Brief Title: Testing Use of Condoms on Regression of Cervical Intraepithelial Neoplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Hospital - and gynaecological out-patient clinics in Central Region Denmark (Unknown); Hospital - and gynaecological out-patient clinics in Region Zealand (Unknown); Research grant from Fonden for Faglig Udvikling af Speciallægepraksis (Unknown); Research grant from Kræftens Bekæmpelse (Unknown); Sponsorship for condoms from RFSU (Unknown)
Responsible Party: Principal Investigator, Malene Skorstengaard, MD, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 102-2880/15-3000
Record Dates: First submitted 2016-09-14; First posted 2016-09-20 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: Condom use; Human Papillomavirus; Conization
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Active Comparator): Women who are advised to use condom during the time period between diagnosis and follow-up
  Interventions: Behavioral: Advice to use condoms
- Control group (No Intervention): Women who are not contacted with advise to use condoms

INTERVENTIONS:
Behavioral: Advice to use condoms
  Arms: Intervention group

SUMMARY:
Women who are diagnosed with CIN2 and who have a pregnancy wish are followed up 6 months after the diagnosis with new examinations. The regression rate is based solely on the woman's own ability to clear the cervical lesions. The use of condoms has shown a relatively good protective effect against Human Papillomavirus (HPV) infection. It has furthermore been indicated that condoms increase the regression rate of cervical lesions.

The hypothesis of this study is that the regression rate of cervical intraepithelial neoplasia grade 2 (CIN2) increases when condoms are used consistently in the follow-up period of 6 months.

DETAILED DESCRIPTION:
Use of condoms has shown a considerable protective effect, when used correctly and consistently, against several sexually transmitted infections (STI), including HIV virus, trichomoniasis, chlamydia, and gonorrhea. It has been indicated that use of condoms also offers a relatively good protection against HPV infections. It is furthermore indicated that use of condoms in women with CIN may increase the regression rate of these lesions.

The aim of this randomized controlled trial is to determine if advising women to use condoms during the follow-up period after a CIN2 diagnosis will increase the regression rate. The advice is based on the presumption that condom use will prevent HPV-infection and reinfection to some extent and thereby allow the immune system to clear the HPV-infection and "repair" the CIN-lesion. Based on the literature, we expect regression in non-condom users to be around 22% and regression in condom-users to be 2.5 times larger.

The clinical trial will be conducted as a randomized non-blinded controlled trial. The study will be conducted at hospital- and gynecological outpatient clinics in Central Region Denmark and Region Zealand.

The gynaecologists will obtain oral and written consent from women with an abnormal cytology to allow the project physician to contact them by telephone. The written consent will be compared to a list from the national pathology register for all diagnosed CIN2 in the relevant regions. If there is a match between the two documents, the gynecologists will be contacted to find out if the woman has been informed about the biopsy result and a follow-up after 6 months has been decided. If this is the case, the woman will be included in the study and randomized.

We expect 700 women to be randomized into an intervention- and a control arm. Women in the intervention arm will receive information about the project by telephone by the project physician. The intervention arm will thereafter be subdivided into a condom group and a non-condom group based on the women's acceptance of the intervention. Women in the condom group will be provided with free condoms for the entire study period. The project physician will not contact women in the control group.

From the routine samples taken at the first visit and at the follow-up examination, an HPV test will be requested from the pathology departments for the women in the condom group. The women are also asked to fill out a questionnaire at the follow-up. The information from the questionnaire is used to estimate compliance to the condom use and to have background information about the women in the condom group.

The study is approved by the Data Protection Agency and the Ethical Committee of the Capital Region of Denmark. The total period of time in which the trial is planned to include women is one year having the last woman to her follow-up visit 18 months after the beginning of the trial. The inclusion period is expected to commence 15.09.16 and end 15.09.17.

Randomization will be conducted electronically by the statistician of the department but neither the investigator nor the patient will be blinded as it is not possible for this study design. Data for the study will be collected from registers and from the questionnaires. All final results from the study will be published in relevant international journals.

The project is supported by funds and we have received a sponsorship for condoms. The sponsors had no influence on the study design, and will have no influence on the data collection, analysis and reporting.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women with CIN2 diagnosed at colposcopy, biopsy and cytology by participating gynaecologist and pathologists and for whom it has been decided to follow-up 6 months later with new examinations at the gynaecologist.

Exclusion Criteria:

* Women with latex allergy
* Women who become pregnant in the study period

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 285 (Actual)
Dates: Start 2016-09; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Regression rate in cervical intraepithelial neoplasia | 6 months follow-up period (The follow-up period at the gynaecologist after the diagnosis of CIN2)
  Difference in regression of CIN2 between the intervention- and control group. Regression is defined as less than CIN2 diagnosis at the 6 months follow-up. For the primary outcome an intention-to-treat analysis will be performed when comparing the intervention group with the control group. Furthermore two per-protocol analysis will be performed. One defining the per-protocol group as those who agreed to use condoms and one defining the per-protocol group who retrospectively reported to use the condoms. Both analysis will be made with control for selection bias.

SECONDARY OUTCOMES:
HPV-clearance | 6 months follow-up period (The follow-up period at the gynaecologist after the diagnosis of CIN2)
  High-risk HPV clearance (type 16,18 or other high-risk types) in the condom user group. Clearance is defined as no high-risk HPV at the 6 months follow-up. Association between CIN2 regression and high-risk HPV clearance will be analysed.

OTHER OUTCOMES:
Questionnaire | 6 months follow-up period (The follow-up period at the gynaecologist after the diagnosis of CIN2)
  The questionnaire variables as predictors of CIN2 regression and as predictors of high-risk HPV clearance.

CONTACTS AND LOCATIONS:
Overall Officials: Elsebeth Lynge, Professor, Study Director — University of Copenhagen
Locations (1):
- Center of Epidemiology and Screening, Copenhagen, Øster Farimagsgade 5, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Skorstengaard M, Suhr J, Lynge E. Condom use to enhance regression of cervical intraepithelial neoplasia: study protocol for a randomized controlled trial. Trials. 2019 Aug 2;20(1):473. doi: 10.1186/s13063-019-3564-4. PMID 31375148